CLINICAL TRIAL: NCT04639830
Title: Electrophysiologic Sleep Phenotyping and Sleep-Dependent Neuro-maturation in Clinical and Healthy Pediatric Populations
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200166; 20-M-0166
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-26

CONDITIONS: Healthy Children; Children With Neurodevelopmental Disorders; Children With Neuropsychiatric Disorders; Children With Behavioral Syndromes
Keywords: SLEEP STUDY; Healthy Children; Neurogenetic Syndrome; Abnormal Neurodevelopment; EEG; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with a known risk: Children between 6 months and 76 months who are at risk for developing a neurodevelopmental disorder.
- Children with no known risk: Children between 6 months and 76 months who don't have a risk for neurodevelopmental disorders.

SUMMARY:
Background:

During the first few decades of life, the brain changes dramatically in shape and function. Sleep lets researchers measure these changes. Researchers want to create a database of sleep and neurodevelopmental data in a group of infants and children to learn more.

Objective:

To address a knowledge and data gap in the field of sleep and neurodevelopment in infants and children.

Eligibility:

Children ages 6 months to 76 months who may or may not be at risk for neurodevelopmental and neuropsychiatric disorders. Also, children ages 6 months to 8 years who have a referral for a sleep study.

Design:

Participants will have neurodevelopmental testing. They will have a medical, psychiatric, and family history. They will have a physical and neurological exam. They will be interviewed and complete surveys. They will give a cheek swab and/or blood sample.

Some participants will have 1 study visit that lasts 2 days.

Other participants will have up to 4 study visits. Each visit will last 2 days. Visits occur every 8 months to 1 year, for a total participation time of 2 years.

Participants will have a 20-minute daytime electroencephalogram (EEG), if possible. This EEG session will be used to calibrate the machine for the overnight study.

Participants will take part in an inpatient overnight sleep study. Electrodes will be placed on the participants. For young children, parents will help place the EEG leads. Other sensors may also be placed. A gauze cap will be placed on participants head to protect the leads and keep the participants from moving them. 'Lights out' will occur as close to participants bedtime as possible.

...

DETAILED DESCRIPTION:
This is a multisite longitudinal study with NIH as the lead site. The other sites: Texas Children s Hospital, Boston Children s Hospital, Geisinger Medical Center, NYU and the NHLBI- supported, area specific repository, National Sleep Research Repository (NSRR). This study will address the data gap established by two NIMH sponsored intramural/extramural workshops (2017 and 2018) in the field of sleep and neurodevelopment by establishing a standardized, reliable protocol for real time acquisition of research data on the normal and abnormal neuro-maturational changes that are sleep-dependent. It will facilitate data-sharing in this area and speed the pace of discovery. Sleep EEG is a highly advantageous modality to provide non-invasive, reliable, robust and reproducible imaging of the brain in young and neurodevelopmentally disordered populations. Sleep EEG affords data acquisition of functional network microstructure with a decreased signal to noise ratio compared to acquisition in the awake state. In addition, potential deviations from the natural ultradian and other sleep oscillatory patterns of the sleep process have the potential to inform on underlying developing neuropathology of various microstructures and neurotransmitter systems prior to the emergence of putatively associated behavioral phenomenon. Ideally, these oscillatory trajectories will not only map to developmental behavioral phenotypes but also to clinical disorders of the sleep state itself, such as the malignant insomnias that are prevalent in neuropsychiatric and neurodevelopmental syndromes. The protocol will initiate the establishment of a normative database for electrophysiologic sleep data in the developing brain. Disorders of particular interest include autism, disorders of social cognition and other neurodevelopmental disorders, childhood psychiatric disorders, and unique clinical presentations of neurogenetic syndromes, such as those associated with genetic disorders or those with a unique family history. The study plans to use a quantitative, dimensional approach to outcome measurement with respect to adaptive functioning in children and to symptoms of behavioral and/or neurodevelopmental problems, irrespective of diagnosis.

While specific differences in the architecture of sleep (e.g., stages, movement abnormalities, cyclicity, spindles and other bio-signatures that reflect anatomical microstructure) may be used to differentiate neurodevelopmental cohorts, the enormous potential of this proposed database lies in the ability to track functional connectivity (coherence) during sleep in the developing brain in a longitudinal, prospective manner, thereby establishing both normal and aberrant trajectories. Predictive relationships can be determined once these trajectories are established. Coherence studies would allow for the potential recreation of neural circuits that sub-serve various brain functions, such as language and attention. Tracking the trajectory of neural development prior to and during the developmental window when these circuits are maturing will allow for an understanding of best potential windows of intervention.

Objectives: The long term, primary objective of this protocol is to evaluate the degree to which the development and maturation of sleep patterns, with an emphasis on the relationship of those patterns to electrophysiologic signals, can predict cognitive and behavioral outcomes. Assessing participants over time will allow researchers to gain additional knowledge about the role of abnormal sleep, measured both clinically and by polysomnogram, in various childhood neuropsychiatric/ neurodevelopmental disorders and behavioral syndromes.

Study Population: The total number of participants to be enrolled will be set at N = 244 (6 months to 8 years old) and will include the following:

1. Study 1: N = 90 with no known risk for neurodevelopmental disorders. These include children without identified neurodevelopmental problems who score within age-expected ranges on cognitive and behavioral screeners.
2. Study 2: N = 154 children at risk for or known to have selected neurodevelopmental/neuropsychiatric disorders, based on any one or more of the following criteria:

   1. Enrolled in early intervention
   2. Getting any targeted therapies
   3. Neurodevelopmental or neuropsychiatric disorder
   4. Failed Infant Toddler Checklist (ITC) (ages 6 months 24 months)
   5. Failed the Early Intervention (EI) screener (>24 months)

Design: Study 1 (N = 90) and Study 2 (N = 154) use the same accelerated longitudinal design.

Outcome Measures: The primary outcome measure in Study 1 is sleep spindle activity. Study 2 has an additional primary outcome, the Vineland Adaptive Behavior (VABS) Socialization growth scale. In both studies, secondary outcome measures will include:other characteristics of sleep spindles, sleep rhythms (ultradian, circadian), macroarchitecture (stages and latencies), microarchitecture (measures of connectivity and network analyses).

Predictors include other neurodevelopmental variables, including other domain scores from the Vineland, IQ, and quantitative measurement of behavioral problems and social communicative development.

ELIGIBILITY:
* INCLUSION CRITERIA :

Inclusion criteria for Group A (No known risk)

-Consent: Parent/caregiver (legal guardian) can give consent. NIH employees children are eligible to participate with the exception of NIMH employees children.

Comments: Parents will provide consent for all minors. Verbal assent will be obtained from minors 7 years and older when applicable.

* The child is between 6 months & 76 months at the time of enrollment for the main study.

Comments: Prescreening assessment

-Apnea hypopnea index (AHI) < 2/hour and no other evidence of sleep disordered breathing (SDB)

Inclusion criteria for Group B (Known risk)

-Consent: Parent/caregiver (legal guardian) can give consent. NIH employees children are eligible to participate with the exception of NIMH employees children.

Comments: Parents will provide consent for all minors. Verbal assent will be obtained from minors 7 years and older when applicable.

-The child is between 6 months & 76 months at the time of enrollment for the main study.

Comments: Screening assessment

-The child meets any one or more of the following:

1. Enrolled in early intervention
2. Getting any targeted therapies
3. Neurodevelopmental or neuropsychiatric disorder
4. Failed ITC (ages 6 months - 24 months)
5. Failed the EI screener (>24 months)
6. Child s first degree relative has been diagnosed with a neurodevelopmental disorder, such as autism or schizophrenia, or severe mental illness, such as major depressive disorder or bipolar disorder

   Comments: Screening assessment
   * Apnea hypopnea index (AHI) <= 2/hour and no other evidence of sleep disordered breathing (SDB)

   EXCLUSION CRITERIA:

   Exclusion criteria for Group A (No known risk)

   -Meets inclusion criteria for Group B (known risk)

   Comments: Screening assessment

   -Any chronic or acute medical condition severe enough to interfere with overnight sleep study acquisition, such as a tracheotomy, uncontrolled seizure disorder, or ventilator dependency, or history of stroke or major neurologic insult. Taking any medications that is known to change sleep parameters within 2 weeks of screening polysomnogram.

   Comments: Screening assessment: Medical history

   -Any history of early intervention or diagnosis of a condition that put the child at risk for neurodevelopmental problems (e.g., genetic disorder, prenatal exposures, extreme prematurity)

   Screening assessment: Medical history

   Primary language other than English in the home

   Comments: Screening assessment

   -Apnea hypopnea index (AHI) >2/hr or any other evidence of sleep disordered breathing (SDB)
   * The children of NIMH employees and staff may not take part.

   Comments: Screening assessment

   Exclusion criteria for Group B (Known risk)

   -Any chronic or acute medical condition severe enough to interfere with completion overnight sleep study acquisition, such as a tracheotomy, uncontrolled seizure disorder, or ventilator dependency.

   Comments: Screening assessment: Medical history

   -Primary language other than English in the home

   Comments: Screening assessment

   -Diagnosed with any of the following common genetic disorders associated with intellectual impairment: Fragile X, Down Syndrome, PraderWilli, Rett, Angelman, Phelan -McDermid, Smith-Lemli-Opitz, identified with a disorders of autonomic dysfunction that might compromise breathing function (examples include congenital central hypoventilation syndrome, familial dysautonmia), disorders of skeletal deformities (Marfan, achondroplasia), a neurogenic condition (spinal muscular atrophy, Duchenne muscular dystrophy, myotonic dystrophy), congenital myopathies or storage diseases (mucopolysaccharidosis, NCL, Wilsons, etc.)

   -The children of NIMH employees and staff may not take part.

   Comments: Screening assessment

   -Apnea hypopnea index > 2/hr or any other evidence of sleep disordered breathing (SDB)

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study Population: The total number of participants to be enrolled will be set at N = 244 (6 months to 8 years old) and will include the following: 1) Study 1: N = 90 with no known risk for neurodevelopmental disorders. These include children without identified neurodevelopmental problems who score within age-expected ranges on cognitive and behavioral screeners. 2) Study 2: N = 154 children at risk for or known to have selected neurodevelopmental/neuropsychiatric disorders, based on any one or more of the following criteria: a) Enrolled in early intervention b) Getting any targeted therapies c) Neurodevelopmental or neuropsychiatric disorder d) Failed Infant Toddler Checklist (ITC) (ages 6 months 24 months) e) Failed the Early Intervention (EI) screener (>24 months)
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Sleep Spindle Activity | ongoing
  The primary outcome measure in Study 1 is sleep spindle activity. Study 2 has an additional primary outcome, the Vineland Adaptive Behavior (VABS) Socialization growth scale.
Vineland Adaptive Behavior (VABS) Socialization growth scale. | ongoing
  The primary outcome measure in Study 1 is sleep spindle activity. Study 2 has an additional primary outcome, the Vineland Adaptive Behavior (VABS) Socialization growth scale.

SECONDARY OUTCOMES:
Sleep Spindle Characteristics | ongoing
  Secondary outcome measures will include: other characteristics of sleep spindles, sleep rhythms (ultradian, circadian), macroarchitecture (stages and latencies), microarchitecture (measures of connectivity and network analyses).

CONTACTS AND LOCATIONS:
Overall Officials: Ashura W Buckley, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (5):
- United States (5):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - New York University - Langone Medical Center, New York, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will use the National Sleep Research Resource (NSRR), based at Brigham and Women s Hospital, as a comprehensive data repository for the visualization, query, and analysis of sleep EEG and related physiologic parameters, neurodevelopmental and demographic data. Most medical and sleep data will be stored using NSRR. All data shared with NSRR will be coded. Samples and data for genomic analyses will be shared with Baylor College of Medicine and they will also be shared with the NIMH Repository & Genomics Resource (NRGR). Coded data from this study for all child participants will also be submitted to the NIH sponsored National Database for Autism Research (NDAR). Data and samples may also be shared with collaborating laboratories at NIH or outside of NIH and/or submitted to NIH-designated repositories and databases if consent for sharing was obtained. Repositories receiving data and/or samples from this protocol may be open-access or restricted access.
Supporting Information: SAP, CSR
Time Frame: IPD and additional supporting information will become available in accordance with the NSRR s and NDAR's policies on public release of data. For other measures, it'll be up to 12 months after the project end date or at the time of acceptance of initial publication, whichever occurs first.
Access Criteria: All data shared with NSRR will be coded; the key to the code will not be provided to collaborators but will remain at NIH. A subset of data shared with NSRR will be stripped of identity and be publicly available. NSRR will initially limit access to only ESP investigators; as the research progresses and with approval from the Steering Committee, de-identified data may be made available to individuals completing appropriate DAUAs.@@@@@@@@@@@@This study will comply with the NIH Genomic Data Sharing Policy, and samples and data for genomic analyses will be shared with Baylor College of Medicine and the NIMH Repository & Genomics Resource (NRGR).@@@@@@@@@@@@Coded data from this study for all child participants will also be submitted to the NIH sponsored National Database for Autism Research, according to NDAR's data sharing policy (which may be found at http://ndar.nih.gov/ndarpublicweb/Documents/NDAR_Policy.pdf).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-M-0166.html